CLINICAL TRIAL: NCT05775965
Title: HIP Fracture Oral ThromboPROphylaxis: a Pilot Randomized Controlled Trial (Hip PRO Pilot)
Brief Title: HIP Fracture Oral ThromboPROphylaxis (Hip PRO Pilot)
Acronym: HIP PRO Pilot
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB22-1085
Record Dates: First submitted 2023-02-07; First posted 2023-03-20 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-09

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Rivaroxaban; Aspirin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban 10mg (Experimental): Rivaroxaban 10mg daily for 35 days post hip fracture surgery
  Interventions: Drug: Rivaroxaban 10mg
- acetylsalicylic acid (ASA) 81mg daily (Experimental): acetylsalicylic acid (ASA) 81mg daily for 35 days post hip fracture surgery
  Interventions: Drug: acetylsalicylic acid (ASA) 81mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 10mg — Rivaroxaban 10mg daily for 35 days post hip fracture surgery
  Other Names: Rivaroxaban
  Arms: Rivaroxaban 10mg
Drug: acetylsalicylic acid (ASA) 81mg Oral Tablet — acetylsalicylic acid (ASA) 81mg daily for 35 days post hip fracture surgery
  Other Names: Aspirin
  Arms: acetylsalicylic acid (ASA) 81mg daily

SUMMARY:
As our Canadian population ages, hip fractures in these older adults are becoming very common. The best treatment for the majority of these injuries is urgent treatment with surgery. However, the hip fracture itself, the surgery required, and the immobility following these injuries are all risk factors for developing blood clots in the legs (deep vein thrombosis or DVT) and blood clots in the lungs (pulmonary embolism or PE). These complications are a common cause of death in patients with hip fractures and often result in prolonged medical treatment and hospital stays.

Patients with hip fractures who require surgery are traditionally given injectable blood thinners to help prevent blood clots; however, these medications are costly, may not be tolerated well, and can be difficult to take, as prescribed. Oral blood thinning medications are being used more commonly, but it is unknown which of these medications is the most effective in preventing blood clots in patients after a hip fracture.

Thrombelastography (TEG) technology uses a small sample of blood to evaluate a person's clotting ability. Our research has used TEG technology to evaluate blood clotting risk after hip fracture surgery and the investigators have found that platelets may play an important role in abnormal blood clotting after a hip fracture. The investigators have also shown that acetylsalicylic acid (ASA or Aspirin) may help reduce the abnormal platelet hyperactivity associated with blood clotting. This medication warrants investigation for blood clot prevention after hip fracture.

The investigators propose to directly compare different oral medication regimens after hip fracture surgery, in order to determine which is safest and most effective in preventing blood clots. Our multi-disciplinary research team includes physicians, surgeons, and scientists with experience evaluating different medications for blood clot prevention. Our results will help determine the best medical treatment for preventing DVT and PE, which will benefit patients with hip fractures worldwide.

DETAILED DESCRIPTION:
1. Background:

   With over 30,000 hip fractures in Canada annually, these injuries are an epidemic. Venous thromboembolism (VTE) events are common following hip fracture surgery (HFS) and include life-threatening pulmonary embolism (PE; a leading cause of preventable mortality) and debilitating deep vein thromboses (DVTs; second most common complication). Thromboprophylaxis reduces VTE, but the optimal medication remains unknown.

   Low molecular weight heparin (LMWH) has been the mainstay, but adherence is poor: only 1 in 5 patients adhere after HFS, limiting its effectiveness. Meta-analyses support that direct oral anticoagulants (DOACs) are as effective as LMWH in prevention of VTE, but the data are limited by borderline effect sizes, small sample sizes, and inconsistent outcomes. Our survey found that surgeons report safety concerns and are reluctant to use DOACs due to post-operative bleeding risk.

   Our research demonstrates platelet-dominant hypercoagulability using serial thrombelastography (TEG), reduced platelet activity with aspirin (ASA) use, and maybe increasing comfort with prescribing ASA post-HFS. Randomized controlled trials (RCTs) comparing LMWH and ASA post-injury are limited by non-standardized therapy duration, asymptomatic DVT inclusion, and patient heterogeneity. ASA has been favourably compared to DOACs and LMWH in arthroplasty RCTs examining oral thromboprophylaxis following total hip and total knee arthroplasty. Continued morbidity and mortality, patient and surgeon preference, and our network meta-analysis support the need for comparison between DOAC and ASA for VTE prevention after HFS. Based on our research, our resent network meta-analysis supporting oral thromboprophylaxis, along with patient preference for oral medications, there is a need for comparison between DOAC and ASA for prevention of VTE to reduce the continued morbidity and mortality that ensues following HFS.
2. Objectives:

Specific Aims:

1. Feasibility: This pilot trial will evaluate the feasibility of a full-scale RCT comparing the safety and efficacy of rivaroxaban versus ASA for thromboprophylaxis after HFS, based on achieving recruitment targets, study drug adherence, and participant retention.
2. Safety and Efficacy: Key clinical data will be collected to estimate VTE and bleeding complications to inform the full-scale RCT.

(3) Methods:

This is a multi-centre double-blind pilot trial consisting of consecutive eligible patients 50 years or older requiring HFS who will be randomized (1:1) via web-based randomization to rivaroxaban 10 mg daily for 35 days or ASA 81 mg daily for 35 days, with 90-day follow-up. The primary feasibility outcome measure is an estimate of the mean monthly recruitment rate over 12 months across participating sites, including 95% confidence intervals, with a priori feasibility criteria determining progression to the full trial. Secondary feasibility outcomes are consent and retention rates, and drug adherence.

Secondary clinical outcomes will include symptomatic VTE, major bleeding, clinically relevant non-major bleeding, and 90-day mortality (independently and blindly adjudicated). Intention-to-treat analysis will be used, and subgroup analysis will compare age, sex, gender, and surgical type. Additional patient-reported (the Cumulated Ambulation Score and Clinical Frailty Scale), value-based (direct and indirect costs) and translational (coagulation) outcomes will be included.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 50 years or older with an acute hip fracture (presentation to hospital within 24 hours of injury) that requires surgical treatment will be approached for inclusion in the study:

1. Age ≥ 50 years with a hip fracture (AO-OTA classification 31-A1-A3 and 31-B1-B3) amenable to surgical treatment (presentation to hospital within 24 hours of injury). Patients with additional injuries will be included and any additional injuries will be documented.
2. Both open and closed fractures will be included, and open fractures will be documented.
3. Patients on single agent anti-platelet therapy (i.e., acetylsalicylic acid or clopidogrel) will be included.
4. Signed informed consent or surrogate consent to participate in study.

Exclusion Criteria:

1. Delayed presentation (over 24 hours between hip fracture and presentation to hospital).
2. Pathological fractures secondary to primary cancer or metastatic bone disease.
3. Peri-prosthetic femur fractures.
4. Received more than two doses of any thromboprophylaxis agent post-operatively, prior to randomization.
5. Pre-hospital therapeutic intensity antithrombotic therapy, including LMWH, Warfarin, DOACs, clopidogrel/ticagrelor, or chronic ASA use of any dose in the three months prior to hip fracture.
6. Known inherited bleeding or clotting disorder (factor V Leiden gene mutation, prothrombin gene mutation, protein C or protein S deficiency, antithrombin deficiency).
7. Intracranial hemorrhage requiring serial CT scans of the brain and/or surgical intervention.
8. Contraindication to ASA use (allergy, documented gastrointestinal ulcer within the past year, severe thrombocytopenia [platelet count <50 x109/L at the time of hospital admission]).
9. Contraindication to rivaroxaban use (allergy, acute renal failure [CrCl <30 mL/min]).
10. Participant or surrogate unable to or unwilling to provide consent or complete follow-up. Or surrogate consent not available.
11. Under age 50 years (more likely high energy, multiple injuries).
12. Multiply injured patients who require prolonged thromboprophylaxis or delayed thromboprophylaxis initiation.
13. Patient unable to attend follow-up visits.
14. Currently incarcerated, at a correctional facility.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  Mean number of participants recruited per centre per month, calculated based on the total recruitment

SECONDARY OUTCOMES:
Treatment fidelity | 12 months
  Adherence to study medication and pilot trial protocol
Retention rate | 12 months
  Participant completion of the pilot trial protocol
Consent rates | 12 months
  Consent rates for eligible participants who are approached, including reasons for non-consent
Trial implementation barriers Questionnaire | 12 months
  Trial implementation barriers will be assessed using an implementation barrier questionnaire developed for this study. The questionnaire will include questions about barriers and challenges related to the following: data capture, study management, study team infrastructure, participant-specific, site-specific, intervention, and study design. The implementation barriers will be summarized at the end of the study.
Healthcare cost | 12 months
  Direct and indirect healthcare costs including number of hospital admissions, and number of visits to healthcare providers.
Venous thromboembolism events | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge, 2-week, 4-week, 6-week, 12-week
  Number of venous thromboembolism events
Arterial thromboembolism events | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge, 2-week, 4-week, 6-week, 12-week
  Number of arterial thromboembolism events
Bleeding complications | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge, 2-week, 4-week, 6-week, 12-week
  Major bleeding, clinically relevant non-major bleeding
Mortality | 90 days
  Mortality within 90 days after hip fracture surgery
Frailty | Baseline
  Frailty is measured by Clinical Frailty Scale. A valid tool for evaluating these patients' frailty levels. The score ranges from 1 to 9. The higher scores mean better frailty (worse outcome).
Complete Blood Counts | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge
  Complete Blood Counts
Partial thromboplastin time | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge
  Partial thromboplastin time
activated partial thromboplastin time | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge
  activated partial thromboplastin time
Cumulated Ambulation Score | Baseline and 2 weeks follow up
  A valid tool for evaluating these patients' basic mobility. The score ranges from 0 to 6. The higher scores mean better mobility.
Study Medication Adherence | Baseline, Post-operative day 1, Post-operative day 2, Post-operative day 3, Post-operative day 4, Post-operative day 5, Post-operative day 6, or until hospital discharge, 2-week, 4-week, 6-week, 12-week
  Adherence to study medications

CONTACTS AND LOCATIONS:
Overall Officials: Prism S Schneider, MD, PhD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Columbian Hospital, New Westminster, British Colombia
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No